CLINICAL TRIAL: NCT00825162
Title: A Phase IV, Open Label, Multi-Centre Study to Evaluate the Safety and Tolerability of CSL Limited's Influenza Virus Vaccine in a Paediatric Population Aged >= 6 Months to < 18 Years
Brief Title: Safety Study of CSL Limited's Influenza Virus Vaccine in the Paediatric Population Aged >= 6 Months to < 18 Years
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seqirus (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CSLCT-USF-06-29
Record Dates: First submitted 2009-01-15; First posted 2009-01-19 (Estimated); Results first posted 2011-07-29 (Estimated); Last update posted 2018-05-23 (Actual); Status verified 2018-04

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort A (Experimental): Participants aged 6 months to less than 3 years
  Interventions: Biological: CSL Limited Influenza Virus Vaccine
- Cohort B (Experimental): Participants aged 3 years to less than 9 years
  Interventions: Biological: CSL Limited Influenza Virus Vaccine
- Cohort C (Experimental): Participants aged 9 years to less than 18 years
  Interventions: Biological: CSL Limited Influenza Virus Vaccine

INTERVENTIONS:
Biological: CSL Limited Influenza Virus Vaccine — Single or two-vaccination regimen (0.25mL)
  Arms: Cohort A
Biological: CSL Limited Influenza Virus Vaccine — Single or two-vaccination regimen (0.5mL)
  Arms: Cohort B
Biological: CSL Limited Influenza Virus Vaccine — Single vaccination regimen (0.5mL)
  Arms: Cohort C

SUMMARY:
A Phase IV, Open Label, Multi-Centre Study to Evaluate the Safety and Tolerability Profile of CSL Limited's Influenza Virus Vaccine in a Paediatric Population Aged >= 6 Months to < 18 Years

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female participants aged ≥ 6 months to < 18 years at the time of vaccination;
2. Written informed consent to participate in the study and adherence to all protocol requirements. Consent will be obtained from the participant, parent or guardian as appropriate according to the applicable Independent Ethics Committee (IEC) and local requirements. Participant assent will also be obtained if required by the applicable IEC;
3. Good health, as determined by medical history, and a targeted physical examination;
4. For participants aged < 9 years, born after a normal gestation period (between 36 and 42 weeks);
5. Females of childbearing potential (defined as having experienced their first menstrual cycle) must be abstinent or be using adequate contraceptive precautions e.g. intrauterine contraceptive device, oral contraceptive, or equivalent hormonal contraception (e.g., progestogen-only implant, vaginal contraceptive ring, cutaneous hormonal patch or injectable contraceptives) for at least 2 months after vaccination. Females aged ≥ 9 years must also return a negative urine pregnancy test at enrolment.

Exclusion Criteria:

1. Known hypersensitivity to a previous dose of influenza vaccine or allergy to eggs, chicken protein, neomycin, polymyxin, or any components of the Study Vaccine;
2. Clinical signs of significant active infection and/or an elevated temperature (≥ 38.0°C oral or ≥ 37.5°C axillary) at study entry;
3. Vaccination against influenza virus in the previous 6 months with a seasonal IVV;
4. Vaccination with an experimental IVV (e.g. a candidate pandemic IVV or a novel IVV) in the previous 6 months;
5. Females of child bearing potential, planning to become pregnant or planning to discontinue contraceptive precautions within 2 months of vaccination;
6. Pregnant or lactating females;
7. Clinically significant medical or psychiatric conditions, as follows:

   * For acute conditions (active or recent), the condition required hospitalisation within the last month; or
   * For chronic conditions: the Investigator feels that the chronic condition is unstable, such as illness exacerbations within the previous month:

     i. requiring hospitalisation; ii. with significant organ function deterioration; iii. with major changes to treatment dosages; iv. requiring major new treatments; or
   * The Investigator feels the participant has a clinical condition that may be adversely affected through study participation.
8. Confirmed or suspected immune deficiency (congenital or acquired, including cancer and human immunodeficiency virus infection);
9. History of seizures, with the exception of a past history of a single seizure event at any age more than two years previously;
10. Known history of Guillain-Barré Syndrome;
11. Current treatment with radiotherapy or cytotoxic drugs, or treatment within the 6 months prior to administration of the Study Vaccine;
12. Current (or within the 90 days prior to receiving the Study Vaccine) immunosuppressive or immunomodulative therapy, including systemic corticosteroids, as follows:

    • Chronic or long term corticosteroids: i. Age less than 9 years: ≥ 0.5 mg/kg/day of oral prednisolone or equivalent daily; ii. Age 9 years and above: ≥ 15 mg/day of oral prednisolone or equivalent daily;

    • Sporadic corticosteroids: i. Age less than 9 years: ≥ 1 mg/kg/day of oral prednisolone or equivalent for 2 or more short courses of > 3 days in the 3 months preceding vaccination; ii. Age 9 years and above: ≥ 40 mg/day of oral prednisolone or equivalent for two or more short courses of > 3 days in the 3 months preceding vaccination; Note: Use of topical or inhalant corticosteroids prior to administration of the Study Vaccine or throughout the Study is acceptable
13. Administration of immunoglobulins and/or any blood products within the 3 months preceding the administration of the Study Vaccine or during the study;
14. Current treatment with warfarin or other anticoagulants;
15. Participation in a clinical trial or use of an investigational compound (i.e. a new chemical or biological entity not registered for clinical use) within 90 days prior to receiving the Study Vaccine or entry into such a study during the on study period;
16. Evidence, or history (within the previous 12 months) of drug or alcohol abuse;
17. If, in the Investigator's opinion, the participant should not take part in the clinical study.

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1992 (Actual)
Dates: Start 2009-03; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Lambert, Dr, Principal Investigator — Royal Children's Hospital, Brisbane, Herston, QLD, Australia
Locations (7):
- Australia (7):
  - The Canberra Hospital, Garran, Australian Capital Territory
  - Sydney Children's Clinical Trials Centre, Randwick, New South Wales
  - Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Children's Hospital, Herston, Queensland
  - Women's & Children's Hospital Adelaide, North Adelaide, South Australia
  - Murdoch Children's Research Institute, Melbourne, Victoria
  - Princess Margaret Hospital, Subiaco, Western Australia

REFERENCES:
- [Result] Lambert SB, Chuk LM, Nissen MD, Nolan TM, McVernon J, Booy R, Heron L, Richmond PC, Walls T, Marshall HS, Reynolds GJ, Hartel GF, Hu W, Lai MH. Safety and tolerability of a 2009 trivalent inactivated split-virion influenza vaccine in infants, children and adolescents. Influenza Other Respir Viruses. 2013 Sep;7(5):676-85. doi: 10.1111/irv.12107. Epub 2013 Apr 2. PMID 23551933

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A: Participants aged 6 months to less than 3 years, who received one or two doses of the 2009 Southern Hemisphere formulation of CSL Limited Influenza Virus Vaccine.
- Cohort B: Participants aged 3 to less than 9 years, who received one or two doses of the 2009 Southern Hemisphere formulation of CSL Limited Influenza Virus Vaccine.
- Cohort C: Participants aged 9 to less than 18 years, who received one or two doses of the 2009 Southern Hemisphere formulation of CSL Limited Influenza Virus Vaccine.
Period: Overall Study
Arm/Group | Cohort A | Cohort B | Cohort C
Started | 710 | 880 | 402
Completed | 682 | 859 | 396
Not Completed | 28 | 21 | 6
Not completed — Withdrawal by Subject | 11 | 13 | 3
Not completed — Lost to Follow-up | 9 | 6 | 3
Not completed — Physician Decision | 2 | 0 | 0
Not completed — Move away from the study area | 1 | 0 | 0
Not completed — Unable to attend the study visit | 5 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort B | Cohort C | Total
Number analyzed (Participants) | 710 | 880 | 402 | 1992
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 710 | 880 | 402 | 1992
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 1.84 (0.74) | 5.54 (1.66) | 12.64 (2.48) | 5.66 (4.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 325 | 439 | 202 | 966
  Male | 385 | 441 | 200 | 1026
Region of Enrollment [Number; unit: participants]
  Australia | 710 | 880 | 402 | 1992

OUTCOME MEASURES:

1. Primary Outcome: Frequency and Intensity of Local and Systemic Solicited Adverse Events, Cohort A (6 Months to Less Than 3 Years)
Description: Solicited Local Adverse Events: pain, redness, and swelling/induration. Solicited Systemic Adverse Events: fever, headache, myalgia, nausea/vomiting, diarrhea, loss of appetite, and irritability.
Time Frame: 7 days post-vaccination
Population: The Safety Population comprised all participants who received CSL's IVV and provided at least one safety assessment after vaccination. For the safety analysis of solicited AEs after the second vaccination, only those participants who received a second vaccination and provided safety follow-up after the second vaccination were included.
Measure: Number; unit: Participants
Groups:
- After First Vaccination, Cohort A; After Second Vaccination, Cohort A: Participants aged 6 months to less than 3 years
Arm/Group | After First Vaccination, Cohort A | After Second Vaccination, Cohort A
Number analyzed (Participants) | 703 | 615
Participants
  Any local solicited adverse event | 254 [56.6% to 64.0%] | 167
  Any pain | 160 | 111
  Grade 3 pain | 1 | 2
  Any redness (> 0 mm) | 148 | 109
  Grade 3 redness (> 30 mm) | 2 | 1
  Any swelling / induration (> 0 mm) | 66 | 64
  Grade 3 swelling / induration (> 30 mm) | 2 | 0
  Any systemic solicited adverse event | 424 | 261
  Any fever (≥99.5°F axillary or ≥100.4 °F oral) | 201 | 110
  Grade 3 fever (≥103.1 F°axillary or ≥104 °F oral) | 13 | 6
  Any headache | 25 | 12
  Grade 3 headache (prevent activities) | 1 | 0
  Any myalgia | 26 | 16
  Grade 3 myalgia (prevent activities) | 3 | 1
  Any nausea / vomiting | 79 | 31
  Grade 3 nausea / vomiting (prevent activities) | 12 | 4
  Any diarrhea | 100 | 52
  Grade 3 diarrhea (prevent activities) | 4 | 3
  Any loss of appetite | 141 | 82
  Grade 3 loss of appetite (prevent activities) | 8 | 4
  Any irritability | 295 | 175
  Grade 3 irritability (prevent activities) | 24 | 7

2. Secondary Outcome: Frequency and Intensity of Unsolicited Adverse Events (UAEs)
Description: UAE stands for Unsolicited Adverse Event.
Time Frame: 30 days after each study vaccination
Population: The Safety Population comprised all participants who received CSL's IVV and provided at least one safety assessment after vaccination.
Measure: Number; unit: Participants
Arm/Group | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 703 | 875 | 398
Participants
  Number of participants with at least one UAE | 531 | 521 | 167
  Number of participants reported Grade 1 UAE | 115 | 183 | 63
  Number of participants reported Grade 2 UAE | 300 | 251 | 82
  Number of participants reported Grade 3 UAE | 116 | 87 | 22

3. Primary Outcome: Duration of Local and Systemic Solicited Adverse Events, Cohort A (6 Months to Less Than 3 Years)
Description: as for outcome 1
Time Frame: 7 days post-vaccination
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | After First Vaccination, Cohort A | After Second Vaccination, Cohort A
Number analyzed (Participants) | 703 | 615
Days
  Any pain | 1.83 (1.264) | 1.76 (1.315)
  Any redness (> 0 mm) | 2.55 (1.930) | 2.74 (2.478)
  Any swelling / induration (> 0 mm) | 3.06 (4.011) | 3.20 (3.301)
  Any fever (≥99.5°F axillary or ≥100.4 °F oral) | 1.54 (1.164) | 1.67 (1.148)
  Any headache | 2.50 (4.492) | 1.23 (0.439)
  Any myalgia | 1.54 (1.071) | 1.70 (1.129)
  Any nausea / vomiting | 1.87 (2.587) | 2.84 (4.919)
  Any diarrhea | 2.43 (3.473) | 2.50 (2.573)
  Any loss of appetite | 2.53 (3.204) | 3.02 (4.325)
  Any irritability | 2.28 (2.503) | 2.42 (2.726)

4. Primary Outcome: Frequency and Intensity of Local and Systemic Solicited Adverse Events, Cohort B (3 Years to Less Than 9 Years)
Description: Solicited Local Adverse Events: pain, redness, and swelling/induration. Solicited Systemic Adverse Events: fever, headache, myalgia, nausea/vomiting, diarrhea, and malaise.
Time Frame: 7 days post-vaccination
Population: as for outcome 1
Measure: Number; unit: Participants
Groups:
- After First Vaccination, Cohort B: Participants aged 3 to less than 9 years
- After Second Vaccination, Cohort B: Participants aged 3 Years to Less Than 9 Years
Arm/Group | After First Vaccination, Cohort B | After Second Vaccination, Cohort B
Number analyzed (Participants) | 875 | 634
Participants
  Any local solicited adverse event | 512 | 312
  Any pain | 463 | 282
  Grade 3 pain | 2 | 2
  Any redness (> 0 mm) | 189 | 109
  Grade 3 redness (> 30 mm) | 18 | 7
  Any swelling / induration (> 0 mm) | 137 | 77
  Grade 3 swelling / induration (> 30 mm) | 19 | 8
  Any systemic solicited adverse event | 346 | 157
  Any fever (≥99.5°F axillary or ≥100.4 °F oral) | 171 | 63
  Grade 3 fever (≥103.1 F°axillary or ≥104 °F oral) | 7 | 2
  Any headache | 136 | 38
  Grade 3 headache (prevent activities) | 4 | 4
  Any myalgia | 87 | 34
  Grade 3 myalgia (prevent activities) | 3 | 3
  Any nausea / vomiting | 75 | 35
  Grade 3 nausea / vomiting (prevent activities) | 6 | 5
  Any diarrhea | 40 | 20
  Grade 3 diarrhea (prevent activities) | 2 | 0
  Any malaise | 179 | 72
  Grade 3 malaise (prevent activities) | 14 | 10

5. Primary Outcome: Duration of Local and Systemic Solicited Adverse Events, Cohort B (3 Years to Less Than 9 Years)
Description: as for outcome 4
Time Frame: 7 days post-vaccination
Population: The Safety Population comprised all participants who received CSL's IVV at Visit 1 and provided at least one safety assessment after vaccination. For the safety analysis of solicited AEs after the second vaccination, only those participants who received a second vaccination and provided safety follow-up after the second vaccination were included.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | After First Vaccination, Cohort B | After Second Vaccination, Cohort B
Number analyzed (Participants) | 875 | 634
Days
  Any pain | 1.89 (1.178) | 1.68 (1.030)
  Any redness (> 0 mm) | 2.45 (1.713) | 2.21 (1.316)
  Any swelling / induration (> 0 mm) | 2.48 (1.688) | 2.09 (1.696)
  Any fever (≥99.5°F axillary or ≥100.4 °F oral) | 1.40 (1.114) | 1.58 (1.117)
  Any headache | 1.79 (1.373) | 1.66 (1.311)
  Any myalgia | 1.74 (1.264) | 1.38 (0.590)
  Any nausea / vomiting | 1.52 (1.305) | 1.36 (0.757)
  Any diarrhea | 2.00 (1.593) | 2.00 (1.612)
  Any malaise | 1.89 (1.763) | 2.13 (1.584)

6. Primary Outcome: Frequency and Intensity of Local and Systemic Solicited Adverse Events, Cohort C (9 Years to Less Than 18 Years)
Description: as for outcome 4
Time Frame: 7 days post-vaccination
Population: as for outcome 5
Measure: Number; unit: Participants
Groups:
- Cohort C: Participants aged 9 to less than 18 years
Arm/Group | Cohort C
Number analyzed (Participants) | 398
Participants
  Any local solicited adverse event | 281
  Any pain | 271
  Grade 3 pain | 1
  Any redness (> 0 mm) | 66
  Grade 3 redness (> 30 mm) | 8
  Any swelling / induration (> 0 mm) | 52
  Grade 3 swelling / induration (> 30 mm) | 12
  Any systemic solicited adverse event | 170
  Any fever (≥99.5°F axillary or ≥100.4 °F oral) | 20
  Grade 3 fever (≥103.1 F°axillary or ≥104 °F oral) | 0
  Any headache | 107
  Grade 3 headache (prevent activities) | 2
  Any myalgia | 80
  Grade 3 myalgia (prevent activities) | 0
  Any nausea / vomiting | 21
  Grade 3 nausea / vomiting (prevent activities) | 1
  Any diarrhea | 21
  Grade 3 diarrhea (prevent activities) | 1
  Any malaise | 66
  Grade 3 malaise (prevent activities) | 1

7. Primary Outcome: Duration of Local and Systemic Solicited Adverse Events, Cohort C (9 Years to Less Than 18 Years)
Description: as for outcome 4
Time Frame: 7 days post-vaccination
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Cohort C
Number analyzed (Participants) | 398
Days
  Any pain | 2.02 (1.317)
  Any redness (> 0 mm) | 2.52 (1.867)
  Any swelling / induration (> 0 mm) | 2.81 (1.854)
  Any fever (≥99.5°F axillary or ≥100.4 °F oral) | 1.21 (0.415)
  Any headache | 1.97 (1.851)
  Any myalgia | 2.20 (3.123)
  Any nausea / vomiting | 1.65 (1.164)
  Any diarrhea | 2.23 (1.771)
  Any malaise | 2.56 (1.853)

8. Secondary Outcome: Frequency of Serious Adverse Events
Time Frame: 180 days after the last study vaccination
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 703 | 875 | 398
Participants
  Number of participants with at least one SAE | 19 | 5 | 2
  Number of participants with related SAE | 0 | 0 | 0

9. Secondary Outcome: Frequency of New Onsets of Chronic Illness
Time Frame: 180 days after the last study vaccination
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 703 | 875 | 398
Participants
  Number of participants with at least one NOCI | 10 | 5 | 2
  Number of participants with related NOCI | 2 | 0 | 0

ADVERSE EVENTS:
Time Frame: SAEs were collected up to 180 days after the last study vaccination. Other adverse events were unsolicited adverse events that were collected up to 30 days after the study vaccination.
Description: Other adverse events were unsolicited adverse events that were collected up to 30 days after the study vaccination.
Arm/Group | Cohort A | Cohort B | Cohort C
Serious Adverse Events (participants affected / at risk) | 19/703 | 5/875 | 2/398
Other Adverse Events (participants affected / at risk) | 531/703 | 467/875 | 97/398
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (N=703) | Cohort B (N=875) | Cohort C (N=398)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Croup infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Eczema infected (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Conversion disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pelvi-ureteric obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (N=703) | Cohort B (N=875) | Cohort C (N=398)
Upper respiratory tract infection (Infections and infestations) | 208 (262) | 142 (171) | 33 (37)
Nasopharyngitis (Infections and infestations) | 50 (59) | 39 (46) | 4 (4)
Respiratory tract infection (Infections and infestations) | 37 (41) | 11 (11) | 3 (3)
Headache (Nervous system disorders) | 2 (3) | 31 (38) | 33 (37)
Cough (Respiratory, thoracic and mediastinal disorders) | 80 (97) | 86 (101) | 6 (6)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 90 (111) | 65 (73) | 12 (13)
Teething (Gastrointestinal disorders) | 113 (165) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 46 (53) | 26 (27) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 36 (40) | 10 (10) | 1 (1)
Pyrexia (General disorders) | 76 (95) | 55 (58) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less